CLINICAL TRIAL: NCT00383890
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study Evaluating the Safety and Efficacy of Dexmedetomidine Used for Sedation During Elective Awake Fiberoptic Intubation
Brief Title: A Safety and Efficacy Study of Dexmedetomidine in Patients Requiring Sedation for Elective Awake Fiberoptic Intubation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospira, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 2005-006; NCT00411775 (obsolete NCT alias)
Record Dates: First submitted 2006-10-02; First posted 2006-10-04 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Awake Fiberoptic Intubation
Keywords: American Society of Anesthesiologists (ASA); Mallampati Score; Ramsay Sedation Scale (RSS)
MeSH Terms: interventions — Dexmedetomidine

ARMS (2):
- Dexmedetomidine (Experimental): Dexmedetomidine 1 mcg/kg load for 10 minutes and Dexmedetomidine Maintenance (0.7 mcg/kg/hr) for 15 min
  Interventions: Drug: Dexmedetomidine HCL Injection
- Placebo (PBO) (Placebo Comparator): Placebo load for 10 min and Placebo maintenance for 15 min
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine HCL Injection
  Arms: Dexmedetomidine
Drug: Placebo
  Arms: Placebo (PBO)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of dexmedetomidine versus placebo used for sedation during elective awake fiberoptic intubation.

DETAILED DESCRIPTION:
An awake fiberoptic intubation is indicated for any patient with an anticipated difficult airway because of their anatomy, airway trauma, morbid obesity, or unstable cervical spine injuries. An awake fiberoptic intubation in a non-sedated patient can be extremely stimulating, uncomfortable, and unpleasant. The clinician must focus on maintaining spontaneous breathing, hemodynamic stability, and the patient's comfort. The term "awake" fiberoptic intubation is used to distinguish this procedure from fiberoptic intubations performed under general anesthesia. Although patients may be sedated for "awake" fiberoptic intubation, they need to be responsive and capable of maintaining their own airway without assistance. Vital components of a successful awake fiberoptic intubation include an anesthesiologist experienced in this technique, adequate topicalization of the airway, and a sedated yet cooperative subject.

Benzodiazepines, combined with opioid, are commonly used for anxiolysis and/or analgesia during awake fiberoptic intubations.

Dexmedetomidine has sympatholytic, sedative, analgesic, and anxiolytic effects that attenuate the catecholamine response to perioperative stress. Dexmedetomidine sedates patients by decreasing sympathetic activity and the level of arousal. Further more, dexmedetomidine has been found to facilitate a decrease in salivary secretion, a desirable effect during fiberoptic intubations.

An estimated 100 subjects (50 DEX, 50 PBO) scheduled for an elective awake fiberoptic intubation because of a potentially difficult airway will be randomized prior to intubation at approximately 18 investigative sites.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (≥18 years of age);
2. American Society of Anesthesiologists (ASA) score I - IV inclusive;
3. Male or female. If female, subject is non-lactating and is either:

   1. Not of childbearing potential, defined as post-menopausal for at least 1 year or surgically sterile due to bilateral tubal ligation, bilateral oophorectomy or hysterectomy.
   2. Of childbearing potential but is not pregnant at time of baseline and is practicing one of the following methods of birth control: oral or parenteral contraceptives, double-barrier method, vasectomized partner, or abstinence from sexual intercourse.
4. Requiring awake fiberoptic (oral or nasal) intubation because of anticipated difficult airway. Subjects must meet at least one of the criteria listed below:

   Criteria for Assessing Difficult Airways

   i. History of difficult intubation

   ii. Anticipated difficult airway
   1. Prominent protruding teeth
   2. Small mouth opening
   3. Narrow mandible
   4. Micrognathia
   5. Macroglossia
   6. Short, muscular neck
   7. Very long neck
   8. Limited neck extension
   9. Congenital airway anomalies
   10. Obesity
   11. Known airway pathology
   12. Known airway malignancy
   13. Upper airway obstruction

   iii. Trauma
   1. Face
   2. Upper airway
   3. Cervical spine

   iv. Anticipated difficult mask ventilation

   v. Severe risk of aspiration

   vi. Respiratory failure

   vii. Severe hemodynamic instability
5. Subject (or subject's legally authorized representative) must voluntarily sign and date the informed consent.

Exclusion Criteria:

1. Previous exposure to any experimental drug within 30 days prior to study drug administration;
2. Central nervous system (CNS) disease with an anticipated increased intracranial pressure or cerebrospinal fluid (CSF) leak;
3. Uncontrolled seizure disorder and/or known psychiatric illness that could confound a normal response to sedative treatment;
4. Presence of acute alcohol intoxication;
5. Current (within 14 days of study entry) treatment with an α2-agonist or antagonist;
6. Subject for whom benzodiazepines, dexmedetomidine or other α2-agonists are contraindicated;
7. Subject received an IV or oral (PO) opioid within one hour or intramuscularly within four hours of the start of study drug administration;
8. Subject has acute unstable angina, laboratory confirmed acute myocardial infarction within the past 6 weeks, heart rate <50 bpm, systolic blood pressure (SBP) <90 mmHg, or complete heart block unless they have a pacemaker.
9. Subject has elevated serum glutamic pyruvate aminotransferase/alanine transaminase (SGPT/ALT) and/or Serum glutamic oxaloacetic transaminase/ aspartate aminotransferase (SGOT/AST) values of ≥2 times the upper limit of normal (ULN).
10. Subject has any other condition or factor which, in the Investigator's opinion, might increase the risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2006-08; Primary Completion 2007-01 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
The percentage of subjects requiring rescue midazolam to achieve and/or maintain proper sedation levels throughout the study drug infusion | At baseline and 15 minutes after starting study drug (prior to topicalization), and every 3 minutes thereafter throughout study drug infusion, at the end of topicalization, and prior to administration of any rescue medication.
  Sedation levels (Ramsay Sedation Scale [RSS] score ≥2 [Patient is cooperative, oriented and tranquil])

SECONDARY OUTCOMES:
Total dose of rescue midazolam required to achieve and/or maintain target sedation levels | During the drug maintenance (i.e, Approximately 15 minutes after starting study drug).
Percentage of subjects requiring additional rescue medications other than midazolam to achieve and/or maintain target sedation levels | During the drug maintenance (i.e, Approximately 15 minutes after starting study drug).
Anesthesiologist assessment of ease of subject care | Immediately following discontinuation of study drug, prior to the scheduled surgery/procedure (Approximately 24 hours).
Subject recall and satisfaction assessed 24 hours post study drug | At the end of the 24-Hour Follow-Up Period

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Miami Jackson Memorial Hospital, Miami, Florida
  - University of Illinois Medical Center at Chicago, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Mayo Clinic Rochester, Rochester, Minnesota
  - New York University Medical Center, New York, New York
  - The Mount Sinai School of Medicine, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - VA North Texas Health Care System, Dallas, Texas
  - The University of Texas Medical School at Houston, Houston, Texas
  - The University of Texas, Houston, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - VA Medical Center, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Bergese SD, Candiotti KA, Bokesch PM, Zura A, Wisemandle W, Bekker AY; AWAKE Study Group. A Phase IIIb, randomized, double-blind, placebo-controlled, multicenter study evaluating the safety and efficacy of dexmedetomidine for sedation during awake fiberoptic intubation. Am J Ther. 2010 Nov-Dec;17(6):586-95. doi: 10.1097/MJT.0b013e3181d69072. PMID 20535016